CLINICAL TRIAL: NCT01196091
Title: A Phase 3, Multicenter, Randomized, Double Blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Subcutaneous LY2127399 in Participants With Systemic Lupus Erythematosus (SLE)
Brief Title: A Study of LY2127399 in Participants With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13656; H9B-MC -BCDS (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-09-03; First posted 2010-09-08 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Systemic Lupus Erythematosus; Connective Tissue Disease; Autoimmune Disease
Keywords: Lupus; SLE; Systemic Lupus Erythematosis; autoimmune disease; LY2127399; Immune system disease
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Connective Tissue Diseases; Autoimmune Diseases; Immune System Diseases | interventions — tabalumab; Standard of Care; Anti-Inflammatory Agents, Non-Steroidal; Adrenal Cortex Hormones; Antimalarials; Immunosuppressive Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- LY2127399 every 2 weeks (Experimental): Administered SC
  Interventions: Drug: LY2127399; Drug: Standard of Care
- LY2127399 every 4 wks (Experimental): During the Treatment Period, for blinding purposes, patients will alternate injections of LY2127399 and injections of placebo every 2 weeks.
  Interventions: Drug: LY2127399; Drug: Placebo every 4 weeks; Drug: Standard of Care
- Placebo (Placebo Comparator): Administered SC
  Interventions: Drug: Placebo every 2 weeks; Drug: Standard of Care

INTERVENTIONS:
Drug: LY2127399 — 120 mg administered via subcutaneous (SC) injection for 52 weeks. 240 mg loading dose will be administered as the first dose of study drug.
  Arms: LY2127399 every 2 weeks; LY2127399 every 4 wks
Drug: Placebo every 2 weeks — Administered via subcutaneous injection for 52 weeks. A matching loading dose of corticosteroids, NSAIDs, antimalarials, or immunosuppressants will also be administered at the first dose
  Arms: Placebo
Drug: Placebo every 4 weeks — Administered via subcutaneous injection for 52 weeks.
  Arms: LY2127399 every 4 wks
Drug: Standard of Care
  Other Names: Non-steroidal anti-inflammatory drug; Corticosteroids; Antimalarials (used for SLE); Immunosuppressants

SUMMARY:
The purpose of this SLE study is to evaluate the efficacy, safety and tolerability of two different doses of LY2127399 administered in participants with active SLE.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of SLE by American College of Rheumatology (ACR) criteria
* Have positive antinuclear antibodies (ANA)
* Agree not to become pregnant throughout the course of the trial
* Have a screening SELENA-SLEDAI score ≥6. (The participant must be actively exhibiting all the symptoms scored on the screening SELENA-SLEDAI on the day of screening.)

Exclusion Criteria:

* Have active severe Lupus kidney disease
* Have active Central Nervous System or peripheral neurologic disease
* Have received intravenous immunoglobulin (IVIg) within 180 days of randomization
* Have active or recent infection within 30 days of screening
* Have had a serious infection within 90 days of randomization
* Have evidence or test positive for Hepatitis B
* Have Hepatitis C
* Are human immunodeficiency virus (HIV) positive
* Have evidence of active or latent tuberculosis (TB)
* Presence of significant laboratory abnormalities at screening
* Have had a malignancy in the past 5 years, except for cervical carcinoma in-situ or basal cell or squamous epithelial skin cell that were completely resected with no reoccurrence in the 3 yrs prior to randomization
* Have received greater than 40 mgs of prednisone or equivalent in the past 30 days
* Have changed your dose of antimalarial drug in the past 30 days
* Have changed your dose of immunosuppressive drug in the past 90 days
* Have previously received rituximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1164 (Actual)
Dates: Start 2010-12; Primary Completion 2014-07 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9AM - 5PM Eastern time (UTC/GMT -5 hours, EST), Study Director — Eli Lilly and Company
Locations (192):
- United States (88):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Birmingham, Alabama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glendale, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mesa, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paradise Valley, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peoria, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Phoenix, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Anaheim, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glendale, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lakewood, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Long Beach, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sacramento, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Leandro, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Upland, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Danbury, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Farmington, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Norwich, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trumbull, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boca Raton, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clearwater, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Doral, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Lauderdale, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Mary, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orange Park, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palm Harbor, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., St. Petersburg, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tamarac, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tampa, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Atlanta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Decatur, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marietta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boise, Idaho
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peoria, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Muncie, Indiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kansas City, Kansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bowling Green, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lexington, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hagerstown, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wheaton, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grand Rapids, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Eagan, Minnesota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Florissant, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lincoln, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clifton, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Teaneck, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toms River, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Endwell, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manhasset, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., The Bronx, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Charlotte, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenville, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hickory, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Middleburg Heights, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Edmond, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pittsburgh, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Willow Grove, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Columbia, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Greenville, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., North Charleston, South Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Crossville, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hixon, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jackson, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Allen, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Houston, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Irving, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mesquite, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Antonio, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sugar Land, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waco, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chesapeake, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Danville, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Williamsburg, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tacoma, Washington
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milwaukee, Wisconsin
- Argentina (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Caba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Córdoba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rosario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Miguel de Tucumán
- Austria (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Graz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vienna
- Belarus (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grodno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Minsk
- Bulgaria (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plovdiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sofia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Stara Zagora
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Varna
- Canada (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kelowna, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Markham, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Newmarket, Ontario
- Chile (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osorno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santiago
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Valdivia
- Colombia (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bogotá
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucaramanga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cali
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chía
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Medellín
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osijek, Croatia
- Egypt (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Al Minyā
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alexandria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cairo
- Germany (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Nauheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Baden-Baden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Erlangen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Freiburg im Breisgau
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hildesheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jena
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zerbst
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guatemala City, Guatemala
- Italy (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brescia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Napoli
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Padua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Palermo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Scafati
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torino
- Japan (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aichi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hokkaido
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Japan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miyagi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nagasaki
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
- North Macedonia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bitola
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shtip
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Skopje
- Peru (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arequipa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lima
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lince
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Piura
- Philippines (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Angeles City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cebu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Davao City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ermita
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., España
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Iloilo City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Manila
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paranaque City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Quezon City
- Poland (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., ?Ód?
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bytom
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sosnowiec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroc?Aw
- Puerto Rico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Juan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santurce
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore
- South Korea (8):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucheon-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daegu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Daejeon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gwangju
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Incheon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jeonju
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Suwon
- Thailand (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bangkok
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiang Mai
- Ukraine (13):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Donetsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ivano-Frankivsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kharkiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kryvyi Rih
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyiv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lviv
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Odesa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Simferopol
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ternopil
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Uzhhorod
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vinnytsia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zaporizhzhia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zhytomyr

REFERENCES:
- [Derived] Vendel AC, Jaroszewski L, Linnik MD, Godzik A. B- and T-Lymphocyte Attenuator in Systemic Lupus Erythematosus Disease Pathogenesis. Clin Pharmacol Ther. 2024 Jul;116(1):247-256. doi: 10.1002/cpt.3282. Epub 2024 Apr 26. PMID 38676311
- [Derived] Toro-Dominguez D, Martorell-Marugan J, Martinez-Bueno M, Lopez-Dominguez R, Carnero-Montoro E, Barturen G, Goldman D, Petri M, Carmona-Saez P, Alarcon-Riquelme ME. Scoring personalized molecular portraits identify Systemic Lupus Erythematosus subtypes and predict individualized drug responses, symptomatology and disease progression. Brief Bioinform. 2022 Sep 20;23(5):bbac332. doi: 10.1093/bib/bbac332. PMID 35947992
- [Derived] Li Y, Higgs RE, Hoffman RW, Dow ER, Liu X, Petri M, Wallace DJ, Dorner T, Eastwood BJ, Miller BB, Liu Y. A Bayesian gene network reveals insight into the JAK-STAT pathway in systemic lupus erythematosus. PLoS One. 2019 Dec 2;14(12):e0225651. doi: 10.1371/journal.pone.0225651. eCollection 2019. PMID 31790472
- [Derived] Kalunian KC, Urowitz MB, Isenberg D, Merrill JT, Petri M, Furie RA, Morgan-Cox MA, Taha R, Watts S, Silk M, Linnik MD. Clinical trial parameters that influence outcomes in lupus trials that use the systemic lupus erythematosus responder index. Rheumatology (Oxford). 2018 Jan 1;57(1):125-133. doi: 10.1093/rheumatology/kex368. PMID 29045736
- [Derived] Hoffman RW, Merrill JT, Alarcon-Riquelme MM, Petri M, Dow ER, Nantz E, Nisenbaum LK, Schroeder KM, Komocsar WJ, Perumal NB, Linnik MD, Airey DC, Liu Y, Rocha GV, Higgs RE. Gene Expression and Pharmacodynamic Changes in 1,760 Systemic Lupus Erythematosus Patients From Two Phase III Trials of BAFF Blockade With Tabalumab. Arthritis Rheumatol. 2017 Mar;69(3):643-654. doi: 10.1002/art.39950. PMID 27723281
- [Derived] Rovin BH, Dooley MA, Radhakrishnan J, Ginzler EM, Forrester TD, Anderson PW. The impact of tabalumab on the kidney in systemic lupus erythematosus: results from two phase 3 randomized, clinical trials. Lupus. 2016 Dec;25(14):1597-1601. doi: 10.1177/0961203316650734. Epub 2016 May 24. PMID 27220348
- [Derived] Isenberg DA, Petri M, Kalunian K, Tanaka Y, Urowitz MB, Hoffman RW, Morgan-Cox M, Iikuni N, Silk M, Wallace DJ. Efficacy and safety of subcutaneous tabalumab in patients with systemic lupus erythematosus: results from ILLUMINATE-1, a 52-week, phase III, multicentre, randomised, double-blind, placebo-controlled study. Ann Rheum Dis. 2016 Feb;75(2):323-31. doi: 10.1136/annrheumdis-2015-207653. Epub 2015 Sep 3. PMID 26338095

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Intent to Treat population (ITT) is all randomized participants who received at least 1 dose of study drug, excluding two sites' participants due to good clinical practice (GCP) issues.
Groups:
- LY2127399 Every 2 Weeks: LY2127399: 120 mg administered via subcutaneous injection for 52 weeks. 240 mg loading dose will be administered as the first dose of study drug.
- LY2127399 Every 4 Wks: During the Treatment Period, for blinding purposes, patients will alternate injections of LY2127399 and injections of placebo every 2 weeks.
  LY2127399: 120 mg administered via subcutaneous injection for 52 weeks. 240 mg loading dose will be administered as the first dose of study drug.
  Placebo every 4 weeks: Administered via subcutaneous injection for 52 weeks.
- Placebo: Placebo every 2 weeks: Administered via subcutaneous injection for 52 weeks. A matching loading dose will also be administered at the first dose
Period: Overall Study
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Wks | Placebo
Started | 387 | 389 | 388
Received at Least 1 Dose of Study Drug | 386 | 389 | 387
ITT-Received Drug and Excluded Sites | 381 | 378 | 379
Follow-Up | 103 | 105 | 128
Completed | 299 | 291 | 284
Not Completed | 88 | 98 | 104
Not completed — Adverse Event | 22 | 27 | 26
Not completed — Death | 3 | 2 | 2
Not completed — Entry Criteria Not Met | 11 | 11 | 10
Not completed — Lack of Efficacy | 15 | 12 | 17
Not completed — Lost to Follow-up | 5 | 5 | 6
Not completed — Parent/Caregiver Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 16 | 19 | 22
Not completed — Physician Decision | 3 | 3 | 4
Not completed — Protocol Violation | 1 | 3 | 3
Not completed — Sponsor Decision | 6 | 5 | 4
Not completed — Excluded Site | 5 | 11 | 8
Not completed — Randomized, No Study Drug Received | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent to Treat population (ITT) all randomized participants who received at least 1 dose of study drug: except those at Sites 301 and 383, which were excluded due to suspected good clinical practice (GCP) issues.
Groups:
- Total: Total of all reporting groups
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Wks | Placebo | Total
Number analyzed (Participants) | 381 | 378 | 379 | 1138
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (12.51) | 40.2 (11.21) | 39.1 (11.69) | 39.7 (11.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 354 | 352 | 360 | 1066
  Male | 27 | 26 | 19 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 119 | 116 | 122 | 357
  Not Hispanic or Latino | 233 | 225 | 229 | 687
  Unknown or Not Reported | 29 | 37 | 28 | 94
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 65 | 55 | 67 | 187
  Asian | 68 | 61 | 66 | 195
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 40 | 41 | 39 | 120
  White | 204 | 218 | 205 | 627
  More than one race | 4 | 2 | 2 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Colombia | 16 | 10 | 18 | 44
  Argentina | 20 | 24 | 22 | 66
  Puerto Rico | 3 | 7 | 11 | 21
  Singapore | 0 | 2 | 0 | 2
  United States | 128 | 133 | 116 | 377
  Philippines | 26 | 14 | 22 | 62
  Japan | 15 | 15 | 15 | 45
  Egypt | 19 | 19 | 21 | 59
  Ukraine | 23 | 22 | 29 | 74
  Thailand | 14 | 9 | 11 | 34
  Belarus | 4 | 6 | 2 | 12
  Canada | 2 | 0 | 2 | 4
  Austria | 3 | 3 | 1 | 7
  Macedonia | 3 | 6 | 3 | 12
  Poland | 19 | 16 | 19 | 54
  Guatemala | 13 | 17 | 13 | 43
  South Korea | 11 | 18 | 14 | 43
  Italy | 1 | 7 | 2 | 10
  Bulgaria | 8 | 11 | 12 | 31
  Chile | 8 | 0 | 5 | 13
  Peru | 32 | 33 | 34 | 99
  Germany | 12 | 5 | 7 | 24
  Croatia | 1 | 1 | 0 | 2
Anti-dsDNA Antibody Level [Mean (Standard Deviation); unit: International Units/Milliliter (IU/mL)] | 107.2 (113.50) | 110.4 (111.58) | 107.1 (112.40) | 108.2 (112.41)
Safety of Estrogens in Lupus Erythematosus National Assessment (SELENA-SLEDAI) Score [Mean (Standard Deviation); unit: units on a scale] — Safety of Estrogens in Lupus Erythematosus National Assessment - SLE Disease Activity Index (SELENA-SLEDAI) score is a weighted, cumulative index of lupus disease activity. SELENA-SLEDAI is calculated from 24 individual descriptors across 9 organ systems; 0 indicates inactive disease and the maximum theoretical score is 105.
  units on a scale | 10.2 (3.5) | 10.4 (3.6) | 10.7 (3.9) | 10.4 (3.7)
Physician's Global Assessment (PGA) Score [Mean (Standard Deviation); unit: millimeters (mm)] — PGA is a single-item clinician rated assessment of the participant's current level of disease activity measured on a continuous 0 to 100-millimeter (mm) visual analytic scale with benchmarks of 0, 1, 2, and 3 from left to right corresponding to no, mild, moderate, and severe SLE disease activity. Scores range from 0, being worst possible to 100 being very active or best possible.
  millimeters (mm) | 46.3 (15.7) | 46.1 (16.2) | 47.1 (16.10) | 46.5 (16.0)
Time of Onset of Lupus [Mean (Standard Deviation); unit: years] | 7.5 (7.4) | 8.1 (7.9) | 6.4 (6.8) | 7.3 (7.4)
At Least One BILAG A or Two BILAG B Disease Activity Scores [Count of Participants; unit: Participants] — The British Isles Lupus Assessment Group (BILAG) instrument assesses global disease activity across 9 organ system domains. BILAG flare is assessed for each of the 9 organ domains using BILAG2004 index flare rules; A is a severe flare and B is a moderate flare.
  The sum of participants in all Categories for the Measure does not equal the Overall Number of Baseline Participants in the Arm/Group because not all participants will have at least one BILAG A or Two BILAG B Disease Activity scores.
  Participants
    Yes | 360 | 340 | 347 | 1047
    No | 21 | 38 | 31 | 90
Lupus Quality of Life (lupus QOL) Domain Score [Mean (Standard Deviation); unit: units on a scale] — The LupusQoL is a disease-specific, 34-item, self-report questionnaire designed to measure the health-related quality of life (HRQoL) of participants with SLE within 8 domains.Responses are based on a 5-point Likert scale where 0 (all of the time) to 4 (never). A LupusQoL score for each domain is reported on a 0 to 100 scale, with greater values indicating better HRQoL.
  units on a scale
    Physical Health | 59.2 (24.98) | 59.1 (25.13) | 56.9 (26.17) | 58.4 (25.43)
    Emotional Health | 65.7 (25.19) | 66.7 (23.99) | 64.6 (26.22) | 65.7 (25.14)
    Body Image | 61.1 (28.99) | 63.2 (27.67) | 61.9 (29.20) | 62.1 (28.61)
    Pain | 56.1 (28.40) | 56.9 (26.75) | 53.6 (28.62) | 55.5 (27.95)
    Planning | 61.2 (30.37) | 62.1 (28.69) | 59.0 (30.92) | 60.8 (30.01)
    Fatigue | 56.0 (26.39) | 54.4 (25.54) | 53.4 (27.14) | 54.6 (26.36)
    Intimate Relationships | 56.2 (33.92) | 63.3 (31.53) | 56.8 (34.21) | 58.8 (33.36)
    Burden to Others | 52.8 (30.70) | 51.9 (30.31) | 49.3 (32.39) | 51.3 (31.15)
Brief Fatigue Inventory (BFI) Score (Worst Level of Fatigue in the Last 24 Hours) [Mean (Standard Deviation); unit: units on a scale] — BFI is a participants-reported scale that measures the severity of fatigue based on the worst fatigue experienced during the past 24-hours. The severity scores ranged from 0 (no fatigue) to 10 (fatigue as severe as you can imagine).
  units on a scale | 5.8 (2.57) | 5.6 (2.81) | 5.6 (2.81) | 5.6 (2.73)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving an SLE Responder Index Response at Week 52
Description: Percentage of participants with a ≥ 5 point reduction from baseline in SELENA SLEDAI score, and no worsening (increase of < 0.30 points from baseline) in PGA, and no new BILAG A organ domain score or 2 new BILAG B organ domain scores compared with baseline.
  SELENA SLEDAI is calculated from 24 individual descriptors across 9 organ systems; 0 indicates inactive disease and the maximum theoretical score is 105; scores > 20 are rare. PGA is a visual analog scale scored from 0 to 3 (0=none, 1=mild, 2=moderate, 3=severe). BILAG uses a single score for each of the 9 organ domains; range is from severe (A) to no disease (E). Participants who were unable to comply with allowed concomitant medications requirements were considered non-responders, as were participants who dropped out or were missing Week 52 data.
Time Frame: 52 weeks
Population: Intent to Treat population (ITT) all randomized participants who received at least 1 dose of study drug and evaluable SLE scores, excluding two sites' participants due to good clinical practice (GCP) issues.
Measure: Number; unit: percentage of participants
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Wks | Placebo
Number analyzed (Participants) | 381 | 378 | 379
percentage of participants | 31.8 | 35.2 | 29.3

2. Secondary Outcome: Percentage Participants Able to Decrease Dose of Prednisone or Equivalent With No Increase in Disease Activity at Week 52
Description: A participant achieves corticosteroid sparing effects (quiescent disease) if they have met the following criteria during Weeks 24 through 52; able to decrease their dose of prednisone or equivalent to 7.5 mg/day or less, have quiescent disease (BILAG C score or better in all nine systems), and no BILAG A or B flares in the previous three months, without an increase in either antimalarials or immunosuppressants on or prior to the visit. Only participants receiving a prednisone or equivalent dose of more than 7.5 mg/day at baseline are included.
Time Frame: 52 weeks
Population: All randomized participants who received at least 1 dose of study drug, a baseline use of prednisone or equivalent >7.5 mg/day, excluding two sites' participants due to good clinical practice (GCP) issues.
Measure: Number; unit: percentage of partipants
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Wks | Placebo
Number analyzed (Participants) | 197 | 200 | 196
percentage of partipants | 15.5 | 17.0 | 16.4

3. Secondary Outcome: Change From Baseline to 52 Weeks in Anti-double Stranded Deoxyribonucleic Acid (Anti-dsDNA) Level
Description: Anti-double stranded deoxyribonucleic acid (anti-dsDNA) is a lab analyte used to assist in the diagnosis of SLE.
Time Frame: Baseline, 52 weeks
Population: All randomized participants who received at least 1 dose of study drug, excluding two sites' participants due to good clinical practice (GCP) issues and a non-missing result at Week 52.
Measure: Mean (Standard Deviation); unit: international units
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Wks | Placebo
Number analyzed (Participants) | 381 | 378 | 377
international units | 107.2 (113.50) | 110.4 (111.58) | 107.1 (112.40)

4. Secondary Outcome: Change From Baseline to 52 Week Endpoint in Systemic Lupus Erythematosus Disease Activity Index (SLEDAI2K) Score
Description: SLE Disease Activity Index 2000 (SLEDAI-2K) score is a weighted, cumulative index of lupus disease activity. SLEDAI-2K is calculated from 24 individual descriptors across 9 organ systems; 0 indicates inactive disease and the maximum theoretical score is 105.
Time Frame: Baseline, 52 weeks
Population: All randomized participants who received at least 1 dose of study drug, excluding 2 sites' participants due to GCP issues and non-missing results; LOCF, defined as: endpoint is defined as the latest post-baseline response obtained on or prior to the date of Week 52 or the date of early discontinuation from the treatment period.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Wks | Placebo
Number analyzed (Participants) | 377 | 374 | 376
units on a scale | -4.7 (4.35) | -4.9 (4.32) | -4.6 (4.54)

5. Secondary Outcome: Time to First Severe SLE Flare (SFI)
Description: The SFI uses the SELENA-SLEDAI disease activity index score, disease activity scenarios, treatment changes, and PGA to define mild/moderate and severe flares. The index takes into account the absolute change in total scores, new or worsening symptoms, and increases in corticosteroid use or hospitalization due to the disease activity.
  Time to first severe SLE flare (SFI) (in days) is calculated as: (Start date of first severe SLE flare (SFI) - Date of randomization + 1).
Time Frame: Baseline through 52 weeks
Population: Zero participants analyzed. Time to first severe SLE flare data was not collected for analysis.
Groups:
- Placebo: Placebo every 2 weeks: Administered via subcutaneous injection for 52 weeks. A matching loading dose will also be administered at first dose.
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Wks | Placebo
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Percentage of Participants With No Worsening in Physician Global Assessment (PGA) Score at 52 Weeks
Description: Physician's Global Assessment (PGA) is a single-item clinician rated assessment of the patient's current level of disease activity measured on a continuous 100 millimeter (mm) visual analytic scale with benchmarks of 0, 1, 2, and 3 from left to right corresponding to no, mild, moderate, and severe SLE disease activity. Scores are presented from 0 to 100. No worsening is defined as increase of ≥0.3 points.
Time Frame: 52 weeks
Population: All randomized participants who received at least 1 dose of study drug, excluding two sites' participants due to good clinical practice (GCP) issues
Measure: Number; unit: percentage of participants
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Wks | Placebo
Number analyzed (Participants) | 381 | 378 | 379
percentage of participants | 64.3 | 61.4 | 58.0

7. Secondary Outcome: Change From Baseline to 52 Week Endpoint in Brief Fatigue Inventory (BFI) Scores
Description: A participants-reported scale that measures the severity of fatigue based on the worst fatigue experienced during the past 24-hours. The severity scores ranged from 0 (no fatigue) to 10 (fatigue as severe as you can imagine).
Time Frame: Baseline, 52 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Wks | Placebo
Number analyzed (Participants) | 362 | 363 | 361
units on a scale | -0.9 (3.09) | -0.9 (3.14) | -0.6 (2.86)

8. Secondary Outcome: Change From Baseline to 52 Week Endpoint Lupus Quality of Life (LupusQoL) Domain Scores
Description: The LupusQoL is a disease-specific, 34-item, self-report questionnaire designed to measure the health-related quality of life (HRQoL) of participants with SLE within 8 domains.Responses are based on a 5-point Likert scale where 0 (all of the time) to 4 (never). A LupusQoL score for each domain is reported on a 0 to 100 scale, with greater values indicating better HRQoL.
Time Frame: Baseline, 52 weeks
Population: All randomized participants who received at least 1 dose of study drug, excluding 2 sites' participants due to GCP issues and a non-missing result.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Wks | Placebo
Number analyzed (Participants) | 381 | 378 | 361
units on a scale
  Physical Health: number analyzed (Participants) | 121 | 133 | 111
  Physical Health | 73.7 (26.05) | 72.8 (24.53) | 72.8 (23.70)
  Emotional Health: number analyzed (Participants) | 121 | 133 | 111
  Emotional Health | 75.2 (25.50) | 72.4 (24.08) | 73.1 (25.54)
  Body Language: number analyzed (Participants) | 117 | 131 | 108
  Body Language | 75.1 (26.21) | 75.0 (24.82) | 71.9 (28.90)
  Pain: number analyzed (Participants) | 121 | 133 | 111
  Pain | 74.0 (27.42) | 74.1 (24.94) | 73.2 (27.30)
  Planning: number analyzed (Participants) | 121 | 133 | 111
  Planning | 77.3 (26.53) | 75.0 (29.07) | 74.5 (28.93)
  Fatigue: number analyzed (Participants) | 121 | 133 | 111
  Fatigue | 70.4 (25.51) | 68.8 (26.34) | 64.5 (24.94)
  Intimate Relationships: number analyzed (Participants) | 100 | 124 | 101
  Intimate Relationships | 77.4 (29.01) | 68.8 (34.06) | 68.7 (30.08)
  Burden to Others: number analyzed (Participants) | 121 | 133 | 111
  Burden to Others | 68.7 (30.43) | 63.5 (30.34) | 63.7 (30.21)

9. Secondary Outcome: Time to First New British Isles Lupus Assessment Group (BILAG A) or 2 New BILAG B SLE Flares
Description: The British Isles Lupus Assessment Group (BILAG) instrument assesses global disease activity across 9 organ system domains. BILAG flare is assessed for each of the 9 organ domains using BILAG2004 index flare rules; A is a severe flare and B is a moderate flare.
  Time to first BILAG A or two BILAG B flares (in days) is calculated as: (Start date of first BILAG A or two BILAG B flares - Date of randomization + 1). The two BILAG B flares must occur in different domains at the same visit.
Time Frame: Baseline through 52 weeks
Population: Zero participants analyzed. Time first new British Isles Lupus Assessment Group (BILAG A) or 2 new BILAG B SLE flares data was not collected for analysis.
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Wks | Placebo
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Change From Baseline to 52 Week Endpoint in PGA
Description: Physician's Global Assessment (PGA) is a single-item clinician rated assessment of the patient's current level of disease activity measured on a continuous 100-mm visual analytic scale with benchmarks of 0, 1, 2, and 3 from left to right corresponding to no, mild, moderate, and severe SLE disease activity. Scores range from 0, being worst possible to 100 being very active or best possible.
Time Frame: Baseline, 52 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Wks | Placebo
Number analyzed (Participants) | 375 | 374 | 375
millimeters | -20.8 (21.97) | -20.8 (22.33) | -20.2 (22.42)

11. Secondary Outcome: Percentage of Participants With an Increase in Corticosteroids Dose at 52 Weeks
Description: An increase in corticosteroids at a visit was defined as a change from baseline greater than 2.5 mg/day in dose or prednisone or equivalent using average daily dose of corticosteroids taken since the previous scheduled visit.
Time Frame: 52 weeks
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Wks | Placebo
Number analyzed (Participants) | 381 | 378 | 379
percentage of participants | 6.7 | 9.1 | 8.8

12. Secondary Outcome: Change From Baseline to 52 Weeks Endpoint in SELENA-SLEDAI Disease Activity Score
Description: Safety of Estrogens in Lupus Erythematosus National Assessment - SLE Disease Activity Index (SELENA-SLEDAI) score is a weighted, cumulative index of lupus disease activity. SELENA-SLEDAI is calculated from 24 individual descriptors across 9 organ systems; 0 indicates inactive disease and the maximum theoretical score is 105.
Time Frame: Baseline, 52 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Wks | Placebo
Number analyzed (Participants) | 381 | 378 | 376
units on a scale | -4.6 (4.19) | -4.7 (4.11) | -4.8 (4.47)

13. Secondary Outcome: Percentage of Participants Achieving a Response as Measured by Modified SRI With No BILAG A or No More Than 1 BILAG B Organ Domain Flares at 52 Weeks
Description: Percentage of participants with a ≥ 5 point reduction from baseline in SELENA SLEDAI score, and no worsening (increase of < 0.30 points from baseline) in PGA, and no new BILAG A or no more than 1 new BILAG B organ domain flare compared with baseline. (Primary outcome modified to use BILAG flare instead of BILAG disease score)
  SELENA SLEDAI is calculated from 24 individual descriptors across 9 organ systems; 0 indicates inactive disease and the maximum theoretical score is 105. PGA is a visual analog scale scored from 0 to 3 (0=none, 1=mild, 2=moderate, 3=severe). BILAG flare is assessed for each of the 9 organ domains; A is a severe flare and B is a moderate flare. Patients who were unable to comply with allowed concomitant medications requirements were considered non-responders, as were participants who dropped out or were missing Week 52 data.
Time Frame: 52 weeks
Population: as for outcome 6
Measure: Number; unit: percentage of participants
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Wks | Placebo
Number analyzed (Participants) | 381 | 378 | 379
percentage of participants
  Responder | 31.8 | 35.2 | 29.6
  Non-Responder | 68.2 | 64.8 | 70.4

14. Secondary Outcome: Number of Participants With No New BILAG A and No More Than One New BILAG B Disease Activity Scores Compared to Baseline
Description: The BILAG2004 index is a validated global disease activity index designed on the basis of the physician's ITT, focusing on changes in disease manifestations (new, improved, worsening, etc) occurring in the last 4 weeks compared with the previous 4 weeks.
  The instrument assesses 97 clinical signs, symptoms, and laboratory parameters across 9 organ system domains: constitutional, mucocutaneous, neuropsychiatric, musculoskeletal, cardiorespiratory, gastrointestinal, opthalmic, renal and hematology.
Time Frame: Baseline through 52 weeks
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Wks | Placebo
Number analyzed (Participants) | 381 | 378 | 379
Participants | 247 | 234 | 219

ADVERSE EVENTS:
Description: All participants who received at least 1 dose of study drug.
Groups:
- LY2127399 Every 2 Weeks, Follow Up; LY2127399 Every 4 Wks, Follow Up; Placebo, Follow Up: 24-48 weeks post last dose
Arm/Group | LY2127399 Every 2 Weeks | LY2127399 Every 4 Wks | Placebo | LY2127399 Every 2 Weeks, Follow Up | LY2127399 Every 4 Wks, Follow Up | Placebo, Follow Up
Serious Adverse Events (participants affected / at risk) | 42/386 | 56/389 | 50/387 | 14/103 | 16/105 | 23/128
Other Adverse Events (participants affected / at risk) | 250/386 | 243/389 | 246/387 | 13/103 | 11/105 | 13/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2127399 Every 2 Weeks (N=386) | LY2127399 Every 4 Wks (N=389) | Placebo (N=387) | LY2127399 Every 2 Weeks, Follow Up (N=103) | LY2127399 Every 4 Wks, Follow Up (N=105) | Placebo, Follow Up (N=128)
Antiphospholipid syndrome (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lupus endocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mitral valve prolapse (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sickle cell anaemia with crisis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis atrophic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obstruction gastric (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vasculitis gastrointestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Type III immune complex mediated reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 2 (2) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disseminated tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infected skin ulcer (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mycobacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreas infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 8 (9) | 4 (4) | 0 (0) | 2 (2) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Salpingo-oophoritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Superinfection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 7 (7) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medication error (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SLE arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 5 (5) | 4 (4) | 1 (1) | 2 (3)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Brenner tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Central nervous system inflammation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral venous thrombosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropsychiatric lupus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vasculitis cerebral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Affect lability (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Affective disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glomerulonephritis proliferative (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lupus cystitis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lupus nephritis (Renal and urinary disorders) | 2 (2) | 1 (1) | 4 (4) | 3 (3) | 0 (0) | 7 (7)
Mesangioproliferative glomerulonephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Renal failure chronic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cutaneous lupus erythematosus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Female sterilisation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2127399 Every 2 Weeks (N=386) | LY2127399 Every 4 Wks (N=389) | Placebo (N=387) | LY2127399 Every 2 Weeks, Follow Up (N=103) | LY2127399 Every 4 Wks, Follow Up (N=105) | Placebo, Follow Up (N=128)
Dry eye (Eye disorders) | 8 (8) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 12 (14) | 12 (12) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 10 (11) | 11 (12) | 11 (11) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 11 (11) | 7 (7) | 11 (11) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 22 (26) | 29 (33) | 23 (30) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 8 (9) | 8 (8) | 10 (17) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 12 (13) | 6 (6) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 11 (11) | 7 (7) | 7 (9) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 17 (19) | 31 (42) | 21 (24) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 16 (19) | 14 (17) | 11 (12) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 10 (12) | 15 (16) | 10 (11) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 11 (17) | 7 (10) | 6 (8) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 11 (11) | 8 (9) | 10 (11) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 8 (9) | 10 (14) | 8 (16) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 15 (18) | 19 (19) | 17 (19) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 9 (11) | 8 (10) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 4 (5) | 8 (8) | 9 (10) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 10 (11) | 9 (10) | 11 (12) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 13 (13) | 4 (5) | 9 (9) | 1 (1) | 2 (2) | 3 (3)
Influenza (Infections and infestations) | 9 (10) | 5 (5) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 29 (46) | 33 (35) | 37 (48) | 3 (3) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 6 (7) | 3 (3) | 8 (9) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 13 (17) | 18 (19) | 14 (18) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 16 (22) | 15 (16) | 11 (11) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 55 (86) | 41 (55) | 51 (72) | 3 (3) | 3 (3) | 4 (4)
Urinary tract infection (Infections and infestations) | 68 (100) | 52 (76) | 51 (77) | 6 (6) | 2 (2) | 4 (4)
Vulvovaginal mycotic infection (Infections and infestations) | 7 (7) | 9 (12) | 8 (11) | 0 (0) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 8 (9) | 4 (5) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 9 (11) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (15) | 15 (17) | 11 (14) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (15) | 28 (30) | 19 (24) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 4 (5) | 8 (8) | 7 (7) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (8) | 8 (8) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6) | 10 (12) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (11) | 6 (6) | 9 (9) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (8) | 5 (7) | 8 (9) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 6 (6) | 19 (31) | 15 (15) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 34 (48) | 35 (56) | 45 (54) | 0 (0) | 3 (3) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Anxiety (Psychiatric disorders) | 6 (7) | 8 (8) | 6 (7) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 7 (7) | 12 (13) | 12 (12) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 22 (22) | 17 (17) | 16 (17) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 12 (13) | 18 (18) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 6 (6) | 10 (11) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 14 (14) | 13 (13) | 20 (21) | 4 (4) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to product program termination, not all analyses were completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days